CLINICAL TRIAL: NCT05148832
Title: Association Between Administration of Systemic Corticosteroids and the Recovery of Olfactory and/or Gustatory Functions in Patients With COVID-19: A Prospective Cohort Study
Brief Title: Administration of Systemic Corticosteroids and the Recovery of Gustatory Functions in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Taste COVID-19
Record Dates: First submitted 2021-12-05; First posted 2021-12-08 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Olfactory Dysfunction
Keywords: COVID-19; olfactory dysfunction; Gustatory dysfunction; Corticosteriods
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 67 Covid-19 patients with symptoms of ageusia and anosmia were recruited (that their covid infection was confirmed by using PCR).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cortocosteroid (Experimental): ageusia and anosmia were recruited (that their covid infection was confirmed by using PCR). 10 mg of systemic corticosteroids were prescribed weekly to patients to observe taste and smell sensation recovery. All data were recorded and then analyzed.
  Interventions: Drug: Administration of Systemic Corticosteroid

INTERVENTIONS:
Drug: Administration of Systemic Corticosteroid — 10 mg of systemic corticosteroids were prescribed weekly to patients to observe taste and smell sensation recovery.

SUMMARY:
Coronavirus is a global pandemic with a high mortality rate; it is started in china in 2019 and rapidly spread worldwide, reaching its epidemic peak in March 2020 Coronavirus is a family of viruses that usually affect animals. They also can affect the respiratory system of humans, causing different manifestations such as difficulty in breathing, coughing, fever, invasive lung lesions, and viral pneumonia

DETAILED DESCRIPTION:
Coronavirus is a global pandemic with a high mortality rate; it is started in china in 2019 and rapidly spread worldwide, reaching its epidemic peak in March 2020 Coronavirus is a family of viruses that usually affect animals. They also can affect the respiratory system of humans, causing different manifestations such as difficulty in breathing, coughing, fever, invasive lung lesions, and viral pneumonia Smell and taste dysfunction is more frequent in the initial stages of covid-19 infection that occur within the first five days and may be used as pivotal symptoms in the early diagnosis of the disease

ELIGIBILITY:
Inclusion Criteria:

* all signs and symptoms were recorded included fever >38 °C, fatigue, myalgia, arthralgia, sore throat, headache, and its localization (diffuse, frontal, other localization), rhinorrhea, nasal obstruction, epistaxis, tinnitus, and hearing loss, sneezing, cough, sputum production, hemoptysis, dyspnea, respiratory rate >22, crackling sounds during auscultation, nausea, vomiting, diarrhea, and abdominal pain.

Exclusion Criteria:

* patients with absolute contraindications for systemic corticosteroids administration, pregnant women, smokers, and patients with any systemic disease or taking any medications that cause loss of taste or smell were excluded from this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Taste sensation | 3 months
  recovery of taste sensation by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu B, Guo H, Zhou P, Shi ZL. Characteristics of SARS-CoV-2 and COVID-19. Nat Rev Microbiol. 2021 Mar;19(3):141-154. doi: 10.1038/s41579-020-00459-7. Epub 2020 Oct 6. PMID 33024307
- [Background] Vaira LA, Deiana G, Fois AG, Pirina P, Madeddu G, De Vito A, Babudieri S, Petrocelli M, Serra A, Bussu F, Ligas E, Salzano G, De Riu G. Objective evaluation of anosmia and ageusia in COVID-19 patients: Single-center experience on 72 cases. Head Neck. 2020 Jun;42(6):1252-1258. doi: 10.1002/hed.26204. Epub 2020 Apr 29. PMID 32342566